CLINICAL TRIAL: NCT03805529
Title: Effect of Singing on Endothelial Function and Cardiac Autonomic Regulation
Brief Title: The Singing Heart Study
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jacquelyn Kulinski, Assistant Professor, Medical College of Wisconsin
Other Study IDs: 26191
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2021-09

CONDITIONS: Impact of Singing; Cardiovascular Health; Cardiovascular Risk Factors; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This pilot study will help evaluate the effect of singing on heart rate variability and endothelial function (markers of cardiac health). If study results are positive this will support more research on the use of singing in cardiac rehabilitation.

DETAILED DESCRIPTION:
The intent of this protocol is to evaluate the impact of singing on cardiac hemodynamics and endothelial function, a marker of cardiovascular health and future cardiac risk.

The study is designed to consist of an initial phone screen and 1 index visit. All study-related procedures will be performed by a trained member of the research team. Dr. Kulinski will provide oversight of all study related procedures and will be ultimately responsible for validation of eligibility, and completion of all study-related tasks. Patients in the cardiology clinics at Froedtert Hospital will be made aware of this study by the clinic staff. If interested in participating, the patient will be provided with the study coordinator's phone number and the study team will be provided with the patient's contact information. The study team will first screen the potential subject via a phone conversation.

Once the subject is deemed eligible based on the legibility criteria, they will be mailed a copy of the Institutional Review Board (IRB) consent form to review. If after reviewing information about the study, the potential subject remains interested, a 90-minute visit (with reserved clinic exam room) will be scheduled for the same day as their upcoming clinic appointment (or another day if preferred by the subject). Recruited subjects will be advised to remain fasting (for a minimum of at least 3 hours) until their research study appointment has been completed. They can drink water.

The study subjects will be called from the clinic waiting room at the time of their appointment. The subject will be taken to a quiet clinic exam room for the visit. Phones, beepers and other devices which can cause startling noises should be turned off. restrictive clothing that could interfere with blood flow to the arms will be removed. We will ask the subject to remove watches, rings, or other jewelry on the hands or fingers.

Baseline vital signs (resting heart rate, blood pressure, pulse oximetry), weight and height will be obtained. Blood pressure will be measured from the subject's control arm (dominant arm preferred). The non-dominant arm is recommended as the tested (occluded) arm by the manufacturer. The appropriately-sized (Bluetooth-capable) Heart Rate Variability (HRV) heart rate sensor strap will be applied to the subject as shown (picture). It is recommended to allow 5 minutes to pass between the time of blood pressure measurement and the commencement of the EndoPAT recording. The subject will be asked to refrain from talking. Staff should avoid talking to the subject and between themselves as much as possible. During this time, the blood pressure cuff will be moved to the non-dominant upper arm, and subjects' fingers will be placed into the probes with subject's forearms supported on the arm supports. The index finger is recommended for the study; however, if this finger is unsuitable, a different digit (except the thumb) may be used, so long as the same finger is used on both hands. Written informed consent will be obtained. Subject's positional comfort will be maximized. The subject will be instructed to refrain from moving the fingers to the extent possible.

After 5 minutes since blood pressure was taken, baseline EndoPAT measurements will be obtained. Endo-PAT device will be placed on subjects to measure reactive hyperemia index (RHI) according to a standard protocol (please also see uploaded Endo-PAT manual). Briefly, this includes a stable period of baseline signal recording, followed by rapid inflation of the blood pressure cuff to a supra-systolic level at least 60 mm Hg above systolic blood pressure and no less than 200 mm Hg. Total cessation of blood flow will be verified by total absence of EndoPAT signal from the occluded hand. This occlusion will be maintained for exactly 5 minutes. This may cause mild stress and/or discomfort to the subject, who will be closely monitored. After 5 minutes exactly, the cuff will be completely deflated as quickly as possible. The EndoPAT signal will be recorded for an additional 5 minutes.

The research team member will assist the subject in completing pages 1-4 of the study questionnaire, including demographics, medical history, current medications, current exercise and singing habits and physical limitations and/or mobility issues.

Next, the research team will verify Bluetooth connection to the research iPAD. NO subject information will need to be entered on the iPAD. A 1-minute "pre-singing" baseline HRV measurement will be obtained and recorded (refer to uploaded Data Collection Sheet). An automated blood pressure, heart rate and pulse oximetry will be recorded. A pulse oximetry finger probe will remain in place. In a seated position, the subject will watch and sing along to the 10-minute coaching video that includes a warm-up with vocal exercise and the lyrics to the Star-Spangled Banner, created by co-investigator Tanya Kruse Ruck, DMA, assistant professor of voice at the University of Milwaukee. Approximately 7 minutes into the (10-minute) singing video, a "singing" HRV measurement and automated blood pressure, heart rate and pulse oximetry will be obtained and recorded. The heart rate immediately after singing will be recorded. A "post-singing" HRV measurement will be obtained. After the 1-minute post HRV measurement, the heart rate will be recorded (this will allow us to determine 1-minute heart rate recovery). Another blood pressure and pulse oximetry will be recorded. The pulse oximetry probe will be removed, and the subject's fingers connected to a new set of EndoPAT disposable finger probes.

A second EndoPAT measurement will be started immediately according to the same protocol as above.

The subject will be asked to rate the highest level of exertion while singing, according to the Borg scale. The research team member will record their observation of the subject's singing effort The subject will be asked to complete questions relating to their visit experience.

ELIGIBILITY:
Inclusion Criteria:

* Cardiology clinic patients age ≥ 18, willing and able to sign informed consent
* Fasting for at least 3 hours (by time of research appointment)

Exclusion Criteria:

* Subjects with a permanent pacemaker or implantable cardioverter defibrillator (ICD) implanted
* Patients with a history of atrial fibrillation
* Parkinson's disease or a tremor
* Amputated upper extremity or presence of upper-arm (dialysis) fistula
* Fingernail onychomycosis (fungal infections resulting in thickening of the nails)
* Pregnancy
* Current illicit drug use (marijuana, tobacco, cocaine, amphetamines, etc.)
* Current excessive alcohol use (defined as more than 14 drinks/week for women, more than 28 drinks/week for men)
* Unstable coronary heart disease (active symptoms of chest discomfort)
* Subjects requiring supplemental oxygen use
* Non-english speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology clinic patients age ≥ 18, willing and able to sign informed consent
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
The change in heart rate variability during singing | through study completion, an average of 1 year
  Use a professional singing coach to guide subjects through a 10-minute period of singing
The change from baseline vascular endothelial function in subjects who've participated in singing intervention | Change from baseline endothelial function after 10 minutes of singing
  Measure endothelial function (reactive hyperemia index, RHI) through finger plethysmography using EndoPAT

SECONDARY OUTCOMES:
The change in cardiac hemodynamics | Change from baseline heart rate variability after 10 minutes of singing
  Heart rate variability will be measured before, during and post singing
The change in cardiac hemodynamics | Change from baseline blood pressure variability after 10 minutes of singing
  blood pressure will be measured before, during and post singing
The change in cardiac hemodynamics | Change from baseline heart rate variability after 10 minutes of singing
  Heart rate will be measured before, during and post singing
The change in cardiac hemodynamics | Change from baseline pulse ox. after 10 minutes of singing
  Pulse ox. will be measured before, during and post singing
Asses subjects' self-assessment of perceived exertion during singing | after 10 minutes of singing
  subjects perceived exertion during singing using qualitative Borg Rated Perceived Exertion Scale and correlate with changes in cardiac hemodynamics and heart rate variability. Scale is numerical from 6-20, 6 being no exertion at all and 20 being maximal exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The data may be available to qualified investigators following study completion and initial publication of the data with collaboration with the study PI

REFERENCES:
- [Derived] Somayaji K, Frenkel M, Tabaza L, Visotcky A, Ruck TK, Ofori EK, Widlansky ME, Kulinski J. Acute effects of singing on cardiovascular biomarkers. Front Cardiovasc Med. 2022 Jul 18;9:869104. doi: 10.3389/fcvm.2022.869104. eCollection 2022. PMID 35924212